CLINICAL TRIAL: NCT04538950
Title: PET/CT Quantitative Assessment of Myocardial Blood Flow Changes in Oncologic Patients Receiving Checkpoint Inhibitor Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John P. Bois, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-009189
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Positron Emission Tomography Computed Tomography; Radiopharmaceuticals; Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Checkpoint Inhibitor (ICI) (Other): Subjects diagnosed with cancer and will be receiving immune checkpoint inhibitors as treatment standard of care will have a PET/CT scan before and after therapy. PET/CT scan is done for study purposes only.
  Interventions: Diagnostic Test: PET/CT; Drug: radioactive drug (tracer)

INTERVENTIONS:
Diagnostic Test: PET/CT — Positron emission tomography-computed tomography is an image test that helps show detail about how tissues and organs are functioning.
Drug: radioactive drug (tracer) — A radioactive drug (tracer) is used in the PET scan.

SUMMARY:
Researchers are trying to determine the side effects on the heart from immune checkpoint inhibitor (ICI) treatment in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* First time administration of ICI
* Willing and able to return in 4-6 weeks for follow-up study
* Patients with previous heart conditions included (while this may impact MFR the delta MFR is what we are assessing)

Exclusion Criteria:

* Age < 18 years
* Women who are pregnant, or breast-feeding.
* Unable or unwilling to give consent to undergo PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bois, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Checkpoint Inhibitor (ICI)
Started | 6
Completed | 2
Not Completed | 4
Not completed — Pulmonary Issues | 2
Not completed — illness | 2

BASELINE CHARACTERISTICS:
Arm/Group | Checkpoint Inhibitor (ICI)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 68.17 [59 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Microvascular Damage/Endothelial Dysfunction
Description: Number of subjects to develop microvascular damage/endothelial dysfunction as determined by the PET/CT scan.
  PET-CT MFR used to assess dynamic changes in MFR that occur pre and post initiation of ICI and thereby potentially identify early cardiotoxicity in patients who might be more prone to more devastating IRAEs such as myocarditis.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Checkpoint Inhibitor (ICI)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 6 weeks on all participants.
Arm/Group | Checkpoint Inhibitor (ICI)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Checkpoint Inhibitor (ICI) (N=6)
Moderate Sepsis (Infections and infestations) | 1 (1)
Mild vomiting (Gastrointestinal disorders) | 1 (1)
Moderate chest pain (Cardiac disorders) | 1 (1)
Mild atrial fibrillation (Cardiac disorders) | 2 (2)
Mild Ileus (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04538950/Prot_SAP_000.pdf